CLINICAL TRIAL: NCT06408753
Title: Plasma Biomarker in Predicting Response and Toxicity in Hepatocellular Carcinoma Patients Treated With Checkpoint Inhibitors With or Without Sterotatic Body Radiotherapy
Brief Title: Plasma Biomarker in Predicting Response and Toxicity in HCC Patients Treated With Checkpoint Inhibitors With or Without SBRT
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Leung Chiang, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 19-857
Record Dates: First submitted 2021-09-09; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Stereotactic Body Radiotherapy
Keywords: SBRT; immune checkpoint inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: sterotatic body radiotherapy — checkpoint inhibitors with or without sterotatic body radiotherapy

SUMMARY:
This is a prospective study to investigate the biomarkers in predicting treatment outcome and toxicity in hepatocellular carcinoma (HCC) patients receiving immune checkpoint inhibitors with or without stereotactic body radiotherapy (SBRT).

ELIGIBILITY:
Inclusion Criteria:

First Cohort (SBRT+IO):

1. Unresectable HCC confirmed by multi-disciplinary team
2. Tumor size 5-15cm
3. Number of lesion(s) ≤ 3
4. No main portal vein or inferior vena cava thrombosis
5. ECOG performance status 0-1
6. Child-Pugh class A-B7
7. Liver volume minus gross tumor volume > 700ml
8. Adequate organ function
9. No prior systemic therapy, immunotherapy, TACE, radiotherapy, or radio-embolization

Second Cohort (IO alone):

1. BCLC stage C HCC
2. ECOG performance status 0-1
3. Child-Pugh class A5-B9
4. Adequate organ function

Exclusion Criteria:

1. Based on the inclusion criteria above. Any eligibility factors that do not fit the inclusion criteria will be considered as ineligible subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the inclusion criteria above. Any eligibility factors that do not fit the inclusion criteria will be considered as ineligible subjects.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Exosomal PD-L1 level in serum | from the date of first study treatment to the date of last study treatment, an average of 3 years
  Increase in level of exosomal PD-L1 may reflect reinvigoration of T-cell activity against cancer cells, thus predicting the treatment efficacy and toxicities in HCC patients received immunotherapy with or without SBRT
Immune profile of peripheral blood mononuclear cells (PBMC) | from the date of first study treatment to the date of last study treatment, an average of 3 years
  Immune profile of pre-treatment peripheral blood is predictive of sustained responder of radio-embolization, thus predicting the treatment efficacy and toxicities in HCC patients received immunotherapy with or without SBRT

SECONDARY OUTCOMES:
Serum Cytokine profile | from the date of first study treatment to the date of last study treatment, an average of 3 years
  SBRT activates the host immune system, in particular those achieving clinical response to the combined treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Background] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Background] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075
- [Background] Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, Kitano S, Mu Z, Rasalan T, Adamow M, Ritter E, Sedrak C, Jungbluth AA, Chua R, Yang AS, Roman RA, Rosner S, Benson B, Allison JP, Lesokhin AM, Gnjatic S, Wolchok JD. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31. doi: 10.1056/NEJMoa1112824. PMID 22397654
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Wu AY, Ueda K, Lai CP. Proteomic Analysis of Extracellular Vesicles for Cancer Diagnostics. Proteomics. 2019 Jan;19(1-2):e1800162. doi: 10.1002/pmic.201800162. Epub 2019 Jan 11. PMID 30334355
- [Background] Yang Y, Li CW, Chan LC, Wei Y, Hsu JM, Xia W, Cha JH, Hou J, Hsu JL, Sun L, Hung MC. Exosomal PD-L1 harbors active defense function to suppress T cell killing of breast cancer cells and promote tumor growth. Cell Res. 2018 Aug;28(8):862-864. doi: 10.1038/s41422-018-0060-4. Epub 2018 Jun 29. No abstract available. PMID 29959401
- [Background] Chen G, Huang AC, Zhang W, Zhang G, Wu M, Xu W, Yu Z, Yang J, Wang B, Sun H, Xia H, Man Q, Zhong W, Antelo LF, Wu B, Xiong X, Liu X, Guan L, Li T, Liu S, Yang R, Lu Y, Dong L, McGettigan S, Somasundaram R, Radhakrishnan R, Mills G, Lu Y, Kim J, Chen YH, Dong H, Zhao Y, Karakousis GC, Mitchell TC, Schuchter LM, Herlyn M, Wherry EJ, Xu X, Guo W. Exosomal PD-L1 contributes to immunosuppression and is associated with anti-PD-1 response. Nature. 2018 Aug;560(7718):382-386. doi: 10.1038/s41586-018-0392-8. Epub 2018 Aug 8. PMID 30089911
- [Background] Engelhardt B, Ransohoff RM. Capture, crawl, cross: the T cell code to breach the blood-brain barriers. Trends Immunol. 2012 Dec;33(12):579-89. doi: 10.1016/j.it.2012.07.004. Epub 2012 Aug 25. PMID 22926201
- [Background] Kunkel EJ, Butcher EC. Chemokines and the tissue-specific migration of lymphocytes. Immunity. 2002 Jan;16(1):1-4. doi: 10.1016/s1074-7613(01)00261-8. PMID 11825560
- [Background] Harlin H, Meng Y, Peterson AC, Zha Y, Tretiakova M, Slingluff C, McKee M, Gajewski TF. Chemokine expression in melanoma metastases associated with CD8+ T-cell recruitment. Cancer Res. 2009 Apr 1;69(7):3077-85. doi: 10.1158/0008-5472.CAN-08-2281. Epub 2009 Mar 17. PMID 19293190
- [Background] Spranger S, Bao R, Gajewski TF. Melanoma-intrinsic beta-catenin signalling prevents anti-tumour immunity. Nature. 2015 Jul 9;523(7559):231-5. doi: 10.1038/nature14404. Epub 2015 May 11. PMID 25970248
- [Background] Zhang ZN, Zhu ML, Chen YH, Fu YJ, Zhang TW, Jiang YJ, Chu ZX, Shang H. Elevation of Tim-3 and PD-1 expression on T cells appears early in HIV infection, and differential Tim-3 and PD-1 expression patterns can be induced by common gamma -chain cytokines. Biomed Res Int. 2015;2015:916936. doi: 10.1155/2015/916936. Epub 2015 Jan 22. PMID 25685816
- [Background] Lim SY, Lee JH, Gide TN, Menzies AM, Guminski A, Carlino MS, Breen EJ, Yang JYH, Ghazanfar S, Kefford RF, Scolyer RA, Long GV, Rizos H. Circulating Cytokines Predict Immune-Related Toxicity in Melanoma Patients Receiving Anti-PD-1-Based Immunotherapy. Clin Cancer Res. 2019 Mar 1;25(5):1557-1563. doi: 10.1158/1078-0432.CCR-18-2795. Epub 2018 Nov 8. PMID 30409824
- [Background] Chew V, Lee YH, Pan L, Nasir NJM, Lim CJ, Chua C, Lai L, Hazirah SN, Lim TKH, Goh BKP, Chung A, Lo RHG, Ng D, Filarca RLF, Albani S, Chow PKH. Immune activation underlies a sustained clinical response to Yttrium-90 radioembolisation in hepatocellular carcinoma. Gut. 2019 Feb;68(2):335-346. doi: 10.1136/gutjnl-2017-315485. Epub 2018 Feb 13. PMID 29440463
- [Background] Bernstein MB, Krishnan S, Hodge JW, Chang JY. Immunotherapy and stereotactic ablative radiotherapy (ISABR): a curative approach? Nat Rev Clin Oncol. 2016 Aug;13(8):516-24. doi: 10.1038/nrclinonc.2016.30. Epub 2016 Mar 8. PMID 26951040
- [Background] Demaria S, Kawashima N, Yang AM, Devitt ML, Babb JS, Allison JP, Formenti SC. Immune-mediated inhibition of metastases after treatment with local radiation and CTLA-4 blockade in a mouse model of breast cancer. Clin Cancer Res. 2005 Jan 15;11(2 Pt 1):728-34. PMID 15701862
- [Background] Dewan MZ, Galloway AE, Kawashima N, Dewyngaert JK, Babb JS, Formenti SC, Demaria S. Fractionated but not single-dose radiotherapy induces an immune-mediated abscopal effect when combined with anti-CTLA-4 antibody. Clin Cancer Res. 2009 Sep 1;15(17):5379-88. doi: 10.1158/1078-0432.CCR-09-0265. Epub 2009 Aug 25. PMID 19706802